CLINICAL TRIAL: NCT02742415
Title: Caring Hand Massage - an Intervention in Cancer Patients Undergoing Chemotherapy in an Outpatient Setting - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Susanne M. Cutshall, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-001790
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cancer patients receiving hand massage (Experimental): Caring Hand massage will be provided to the outpatients undergoing chemotherapy
  Interventions: Behavioral: Caring Hand Massage

INTERVENTIONS:
Behavioral: Caring Hand Massage — Caring Hand Massage is a hand massage therapy program with several steps and techniques.
  Other Names: Hand Massage Therapy Program

SUMMARY:
Since there is a limited amount of evidence on the feasibility and outcomes on the use of hand massage in patients undergoing cancer treatment, the purpose of this study is to evaluate the feasibility and outcomes of hand massage therapy in cancer patients undergoing chemotherapy, and to measure its influence on their symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 - 80
2. Patient receiving treatment on Mayo Clinic's Chemotherapy Outpatient Clinic
3. Able to speak English and complete surveys
4. Able to read, understand and sign inform consent.

Exclusion Criteria:

1. Patient has rash, sores, wounds, incision or other skin conditions on hands
2. Unable to give consent or complete the surveys
3. Already having received previous hand massage
4. Pregnant women. (As verbalized by participant)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Comparison of symptom scores | baseline to 45 minutes.
  We will record the number of patients approached hand massage to those that accept and were able to get a full hand massage during their time in the chemotherapy area

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Cutshall, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes